CLINICAL TRIAL: NCT03845010
Title: Elimination of Ventricular Premature Beats With CaTheter Ablation Versus OPtImal Anti-arrhythmic Drug Treatment
Brief Title: Elimination of VPB With Ablation Versus Anti-arrhythmic Drug Treatment
Acronym: ECTOPIA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maatschap Cardiologie Zwolle (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 10407
Record Dates: First submitted 2019-01-17; First posted 2019-02-19 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2022-07

CONDITIONS: Ventricular Premature Beats
MeSH Terms: conditions — Ventricular Premature Complexes | interventions — Sotalol; Flecainide; Verapamil; Catheter Ablation

STUDY DESIGN:
Intervention Model Description: Randomized trial comparing catheter ablation with two different potent AADs with different engagement mechanisms in a 1:1:1 ratio with a crossover design in the AAD arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sotalol (Active Comparator)
  Interventions: Drug: Sotalol
- Flecainide and verapamil (Active Comparator)
  Interventions: Drug: Flecainide and verapamil
- Catheter ablation (Active Comparator)
  Interventions: Procedure: Catheter ablation

INTERVENTIONS:
Drug: Sotalol — Patients will be titrated to the maximal tolerated dose of sotalol with a targeted dose of 80 thrice daily (TID)
  Arms: Sotalol
Drug: Flecainide and verapamil — Patients will receive maximal tolerated dose of flecainide and verapamil with titration to a maximal dose of 200 mg of flecainide and 240 mg of verapamil per day
  Arms: Flecainide and verapamil
Procedure: Catheter ablation — Patients will undergo VPB/VT ablation using a percutaneous transfemoral approach according to standard clinical routine
  Arms: Catheter ablation

SUMMARY:
The ECTOPIA trial is a randomized, multicenter, clinical trial to assess elimination of ventricular premature beats (VPB) with catheter ablation versus optimal anti-arrhythmic drugs (AAD) treatment with flecainide/verapamil or sotalol.

DETAILED DESCRIPTION:
The ECTOPIA trial is a randomized, multicenter, clinical trial to assess elimination of VPB with catheter ablation versus optimal AAD treatment with flecainide/verapamil or sotalol. Due to the use of different AAD (with and without beta-blocking abilities) the investigators will be able to explore the secondary objectives. Finally, this study will assess safety of ablation of non-RVOT VPBs and long-term treatment with two different AAD.

ELIGIBILITY:
Inclusion Criteria:

* Patients willing and capable to provide written informed consent
* Patients with frequent symptomatic VPB and/or nonsustained VTs with burden ≥ 5% on 24 hour Holter monitor AND
* Absence of structural heart disease (excluded by echocardiogram) AND
* Absence of underlying cardiac ischemia (ruled out by treadmill test, CT coronary arteries, nuclear scintigraphy or coronary angiography) AND
* Patient is considered an acceptable candidate for catheter ablation treatment with a dominant morphology of VPB/VT origin judged by the treating physician.
* For those already undergoing treatment, all antiarrhythmic drugs including digitalis must be discontinued during a 2-week washout period before entry to the study

Exclusion Criteria:

* Age >75 years
* Previous catheter ablation therapy for VPB/VT
* Patients with sustained ventricular tachycardia or cardiac channelopathies (e.g. Catecholaminergic polymorphic ventricular tachycardia (CPVT), long- or short QT syndrome, Brugada syndrome)
* Wolff-parkinson-white (WPW) syndrome
* Use of medication with risk of QTc prolongation (e.g. antidepressant, antiemetic), except for study medication sotalol.
* Left ventricular dysfunction (LV ejection fraction <55%)
* Estimated glomerular filtration rate < 50 ml/min/1.73 m2
* Hepatic impairment defined by a total bilirubin ≥ 2 times the upper limit (ULN) of normal, or alanine aminotransferase (ALAT) or aspartate aminotransferase (ASAT) ≥ 3 times ULN at screening
* Untreated hypo- or hyperthyroidism or electrolyte imbalance
* Untreated obstructive sleep apnea
* Patients with history of myocardial infarction or bypass surgery
* More than grade 1/3 valvular regurgitation and/or significant valve stenosis (moderate or severe)
* Contraindication for any of the antiarrhythmic drugs used in this study
* Enrolment in another clinical study
* Woman currently pregnant or breastfeeding or not using reliable contraceptive measures during fertile age
* Mental or physical inability to participate in the study
* Life expectancy ≤ 12 months

Min Age: 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 22 (Actual)
Dates: Start 2019-02-12 (Actual); Primary Completion 2023-01-17 (Actual); Study Completion 2023-01-17 (Actual)

PRIMARY OUTCOMES:
Successful therapy | After 3 months
  Number of patients reaching succesfull therapy defined as >80% reduction of of VPB/VT burden after 3 months

SECONDARY OUTCOMES:
VPB/VT burden | 3, 6, 12 months after intervention
Change in VPB/VT burden | Before the intervention (baseline) and 3, 6, 12 months after intervention
  Measurement in different subgroups e.g.: males, pre and post-menopausal women
The impact in terms of total Quality of Life | 3, 6, 12 months after intervention compared to baseline (before intervention)
  Use of the University of Toronto AF severity scale (AFSS) questionnaire to measure Quality of Life. The total score range is 0-35. Seven questions in total with a maximum score of 5 points per question.
Association between number of VPB/hour and heart rate (HR)/hour during 24-hours Holter- monitoring | At baseline
  A scatterplot will be made in order to depict the association between the number of VBP/hour and heart rate (HR)/hour during 24-hour Holter-monitoring
Number of pro-arrhythmic effects, (non)-sustained VT or atrial flutter, in AAD arms with frequent visits and use of 24-hour Holter monitoring | 3, 6 and 12 months after intervention
QTc prolongation (sotalol) and QRS broadening (flecainide) with requiring frequent checks with standard ECG and/or treadmill test | 4-6 weeks after first administration of AAD
Complication rate of catheter ablation | Procedure and 3, 6 and 12 months after intervention
  In all patients with special interest to the subgroup of patients with anatomically challenging origin of (non-RVOT) VPB/VTs
Extended evaluation of left ventricular function with transthoracic echo (TTE) (including global longitudinal strain rate measurement) | Baseline, 6 and 12 months after intervention
Absolute and relative difference in VPB/VT burden (%) from baseline, during treatment with sotalol versus treatment with flecainide/verapamil | 3, 6 and 12 months after intervention
Divide patients in three groups depending on HR dependency of VPB/VT and compare absolute and relative difference in VPB/VT burden (%) from baseline, during treatment with sotalol versus treatment with flecainide/verapamil | 3, 6 and 12 months after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Arif Elvan, MD, PhD, Principal Investigator — Isala
Locations (1):
- Isala hospital, Zwolle, Netherlands

IPD SHARING:
Plan to Share IPD: No